CLINICAL TRIAL: NCT05782777
Title: Effect of High-intensity Statin With Ezetimibe COmbination theRapy Versus High-intensity sTatin Monotherapy After Percutaneous Coronary Intervention With Drug-eluting Stents; the ESCORT Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2022-1335
Record Dates: First submitted 2023-01-29; First posted 2023-03-24 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease Requiring Coronary Revascularization With Newer Generation DES Implantation
MeSH Terms: interventions — Ezetimibe

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination therapy group (Experimental): Ezetimibe/high-intensity statin combination therapy
  Interventions: Drug: ezetimibe/high-intensity statin combination therapy (ezetimibe 10mg plus atoravastatin 40mg)
- Statin monotherapy group (Active Comparator): High-intensity statin monotherapy
  Interventions: Drug: high-intensity statin monotherapy (atoravastatin 40mg)

INTERVENTIONS:
Drug: ezetimibe/high-intensity statin combination therapy (ezetimibe 10mg plus atoravastatin 40mg) — The initial dose of lipid-lowering therapy will be ezetimibe 10mg plus atoravastatin 40mg. During follow-up, the dose of ezetimibe 10mg plus atoravastatin 40mg is strongly recommended to be maintained.
  Arms: Combination therapy group
Drug: high-intensity statin monotherapy (atoravastatin 40mg) — The initial dose of lipid-lowering therapy will be atoravastatin 40mg. During follow-up, the dose of atoravastatin 40mg is strongly recommended to be maintained.
  Arms: Statin monotherapy group

SUMMARY:
This study sought to evaluate whether ezetimibe combination to high-intensity statin therapy will have more prominent beneficial effect compared to high-intensity statin monotherapy in patients who underwent coronary revascularization with newer generation drug-eluting stent (DES) implantation. Furthermore, the optimal OCT-based optimal expansion criteria as well as the efficacy and safety of newer generation will be investigated.

DETAILED DESCRIPTION:
All eligible patients who underwent coronary revascularization with newer generation DES implantation will be enrolled according to inclusion/exclusion criteria after voluntary agreement with informed consent. At the time of enrollment, we will stratify the patients according to LDL-cholesterol <100mg/dL, acute coronary syndrome, and DES type, and randomly assign them in two groups according to lipid-lowering therapy with a 1:1 ratio: "Combination therapy group" vs. "Statin monotherapy group". In this study, four types of new generation DES will be used: Orsiro (Biotronik), Firehawk (Microport), Genoss (Genoss) or D+Storm (CGBIO).

In this study, OCT substudy will be performed for the patients with diffuse long lesions requiring total stented length ≥30 mm (targeted for 700 patients in the trial). Corresponding patients will be randomly assigned into two groups according to the OCT-based optimal expansion criteria with a 1:1 ratio: meeting "Absolute expansion" vs. "Relative expansion". The absolute expansion criteria is defined as a minimum stent area (MSA) >4.5mm2, while the relative expansion criteria is defined as achieving an MSA ≥ 80% of the mean reference lumen area or ≥ 100% of the distal reference lumen area. The patients will receive DES implantation under OCT guidance and stent optimization will be performed to satisfy the assigned expansion criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Age 19-85 years
2. Patients who underwent coronary revascularization with newer generation DES implantation

Exclusion Criteria:

1. Allergy or hypersensitive to ezetimibe or statin
2. Active liver disease or persistent unexplained serum AST/ALT elevation more than 2 times the upper limit of normal range
3. History of any adverse drug reaction requiring discontinuation of statin
4. Pregnant women, women with potential childbearing, or lactating women
5. Life expectancy less than 3 years
6. Inability to follow the patient over the period of 1 year after enrollment, as assessed by the investigator
7. Inability to understand or read the informed consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4310 (Estimated)
Dates: Start 2023-04-07 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Clinical efficacy of lipid lowering therapy | Within 3 years after the enrollment
  Composite of all-cause death, myocardial infarction (MI), any coronary revascularization, hospitalization for unstable angina, or nonfatal stroke within 3 years

SECONDARY OUTCOMES:
Proportion of subjects achieving target LDL-cholesterol <55 mg/dL or 70 mg/dL at 6 weeks, 1, 2, and, 3 years | Within 3 years after the enrollment
Rate of cross-over into the non-allocated therapy | Within 3 years after the enrollment
Each component of primary endpoint A. All-cause death (percentage) | Within 3 years after the enrollment
Each component of primary endpoint B. MI (percentage) | Within 3 years after the enrollment
Each component of primary endpoint C. Any coronary revascularization (percentage) | Within 3 years after the enrollment
Each component of primary endpoint D. Hospitalization for unstable angina (percentage) | Within 3 years after the enrollment
Each component of primary endpoint E. Nonfatal-stroke (percentage) | Within 3 years after the enrollment
Cardiac death (percentage) | Within 3 years after the enrollment
Stent thrombosis (percentage) | Within 3 years after the enrollment
Target-vessel revascularization (percentage) | Within 3 years after the enrollment
Target-lesion revascularization (percentage) | Within 3 years after the enrollment
BARC type 2-5 bleeding (percentage) | Within 3 years after the enrollment
BARC type 3-5 bleeding (percentage) | Within 3 years after the enrollment
Patient-oriented composite endpoint which is composite of all-cause death, MI, or any coronary revascularization (percentage) | Within 3 years after the enrollment
Device-oriented composite endpoint which is composite of cardiovascular death, MI, or clinically-driven target-vessel revascularization (percentage) | Within 3 years after the enrollment
Difference in antiplatelet therapy strategy (percentage) | Within 3 years after the enrollment
Difference in high-ischemic risks (percentage) | Within 3 years after the enrollment
Difference in high-bleeding risks (percentage) | Within 3 years after the enrollment
different OCT optimization criteria when treating very long lesions | Within 3 years after the enrollment
  A. Primary endpoint (percentage) B. Stent thrombosis (percentage) C. Target-vessel revascularization (percentage) D. Target-lesion revascularization (percentage) E. Patient-oriented composite endpoint (percentage) F. Device-oriented composite endpoint ((percentage)
Safety endpoint related to lipid-lowering medication | Within 3 years after the enrollment
  A. New-onset DM, worsening of glycemic control or HOMA-index (percentage) B. Occurrence of SAMS requiring change of therapy regimen or dosage (percentage) C. Elevation of muscle enzymes which is creatine kinase > 4 x Upper Normal Limit (percentage) D. Elevation of hepatic enzymes which is aminotransferase > 3 x Upper Normal Limit (percentage) E. Elevation of serum creatinine level which is > 50% from baseline (percentage) F. Increase of proteinuria (percentage) G. Diagnosis of cancer (percentage)

CONTACTS AND LOCATIONS:
Overall Officials: Byeong-Keuk Kim, Principal Investigator — Severance Cardiovascular Hospital, Yonsei University Health System
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No